CLINICAL TRIAL: NCT06118333
Title: A Phase III Randomized Controlled Trial to Compare BL-B01D1 With Physician's Choice of Chemotherapy (Last Line) in Patients With Recurrent or Metastatic Nasopharyngeal Carcinoma (NPC) Previously Treated With PD-1/PD-L1 Monoclonal Antibody and at Least Two Lines of Chemotherapy (at Least One Line of Platinum-based Chemotherapy)
Brief Title: A Study Comparing BL-B01D1 With Physician's Choice of Chemotherapy in Patients With Recurrent or Metastatic Nasopharyngeal Carcinoma
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sichuan Baili Pharmaceutical Co., Ltd. (Industry)
Collaborators: Baili-Bio (Chengdu) Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BL-B01D1-303
Record Dates: First submitted 2023-10-25; First posted 2023-11-07 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Nasopharyngeal Carcinoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Capecitabine; Gemcitabine; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Participants receive BL-B01D1 as intravenous infusion for the first cycle (3 weeks). Participants with clinical benefit could receive additional treatment for more cycles. The administration will be terminated because of disease progression or intolerable toxicity occurring or other reasons.
  Interventions: Drug: BL-B01D1
- Control group (Experimental): Participants receive capecitabine, gemcitabine, docetaxel in the first cycle (3 weeks). Participants with clinical benefit could receive additional treatment for more cycles. The administration will be terminated because of disease progression or intolerable toxicity occurring or other reasons.
  Interventions: Drug: capecitabine; Drug: gemcitabine; Drug: docetaxel

INTERVENTIONS:
Drug: BL-B01D1 — Administration by intravenous infusion
  Other Names: iza-bren; izalontamab brengitecan; BMS-986507
  Arms: Experimental group
Drug: capecitabine — Oral administration
  Arms: Control group
Drug: gemcitabine — Administration by intravenous infusion
  Arms: Control group
Drug: docetaxel — Administration by intravenous infusion
  Arms: Control group

SUMMARY:
A phase III, randomized, open-label, multicenter study to evaluate the efficacy and safety of BL-B01D1 in patients with recurrent or metastatic nasopharyngeal carcinoma who had failed at least two lines of platinum-based chemotherapy after receiving PD-1/PD-L1 monoclonal antibody as the last line of therapy.

DETAILED DESCRIPTION:
Primary objective: To evaluate BICR-based objective response rate (ORR) and overall survival (OS) benefit of BL-B01D1 versus physician's choice of chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign the informed consent form and comply with the protocol requirements;
2. Age ≥18 years and ≤75 years;
3. Expected survival time ≥3 months;
4. Patients with recurrent or metastatic nasopharyngeal carcinoma confirmed by histology or cytology, who have failed treatment with PD-1/PD-L1 monoclonal antibodies and at least two lines of chemotherapy (including at least one platinum-based regimen);
5. Patients with recurrent or metastatic nasopharyngeal carcinoma suitable for receiving the control group chemotherapy drugs specified in this protocol as the last-line treatment;
6. Must have at least one measurable lesion as defined by RECIST v1.1;
7. ECOG performance status score of 0 or 1;
8. Toxicity from prior anti-tumor treatment has recovered to ≤ Grade 1 as defined by NCI-CTCAE v5.0;
9. No severe cardiac dysfunction, with left ventricular ejection fraction ≥50%;
10. Organ function levels must meet the requirements without transfusion, use of any cell growth factors, and/or platelet-raising drugs within 14 days before randomization;
11. Coagulation function: International Normalized Ratio (INR) ≤1.5, and activated partial thromboplastin time (APTT) ≤1.5×ULN;
12. Urine protein ≤2+ or <1000mg/24h;
13. For premenopausal women with childbearing potential, a serum pregnancy test must be performed within 7 days before starting treatment, and the result must be negative. They must not be breastfeeding. All enrolled patients should take adequate barrier contraception measures throughout the treatment period and for 6 months after treatment ends.

Exclusion Criteria:

1. Use of chemotherapy, targeted therapy, biologic therapy, etc., within 4 weeks or 5 half-lives before randomization, or palliative radiotherapy and antitumor therapy within 2 weeks;
2. Patients with recurrent nasopharyngeal carcinoma suitable for curative-intent local treatment (surgery or radiotherapy) should be excluded;
3. Prior treatment with ADC drugs containing topoisomerase I inhibitor as the small-molecule toxin, or ADC drugs targeting EGFR and/or HER3;
4. History of severe cardiac disease;
5. Unstable thrombotic events requiring therapeutic intervention within 6 months before screening (except for catheter-related thrombosis lasting >4 weeks);
6. QT interval prolongation, complete left bundle branch block, third-degree atrioventricular block, or frequent and uncontrolled arrhythmias;
7. Diagnosis of active malignancy within 3 years before randomization;
8. Poorly controlled hypertension despite two antihypertensive medications, or poorly controlled diabetes, or presence of diabetic gangrene;
9. History of ILD requiring steroid treatment, current ILD, or ≥Grade 2 radiation pneumonitis;
10. Concurrent pulmonary disease resulting in clinically significant respiratory impairment;
11. Imaging findings indicating tumor invasion or encasement of major thoracic, cervical, or vascular structures (if the investigator deems it does not affect patient eligibility, discussion with the sponsor's medical team is required);
12. Patients with active central nervous system metastases;
13. History of allergy to recombinant humanized antibodies or any excipient of BL-B01D1;
14. History of autologous or allogeneic stem cell transplantation;
15. Positive for HIV antibody, active HBV infection, or HCV infection;
16. Severe infection within 4 weeks before randomization, or pulmonary infection or active pulmonary inflammation within 2 weeks before randomization;
17. Pleural effusion, pericardial effusion, or ascites requiring drainage and/or symptomatic within 4 weeks before randomization;
18. Use of other investigational drugs or therapies within 4 weeks before randomization;
19. History of severe neurological or psychiatric disorders;
20. Presence of severe unhealed wounds, ulcers, or fractures within 4 weeks before signing informed consent;
21. Subjects with clinically significant bleeding or obvious bleeding tendency within 4 weeks before signing informed consent;
22. History of intestinal obstruction, inflammatory bowel disease, extensive bowel resection, Crohn's disease, ulcerative colitis, or chronic diarrhea;
23. Subjects planning to receive or having received live vaccines within 28 days before randomization;
24. Any other condition deemed by the investigator to make the patient unsuitable for participation in this clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 386 (Actual)
Dates: Start 2023-12-04 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Up to approximately 24 months
  Objective response rate (ORR) is defined as the number of CR and PR in the treatment and control groups divided by the number of that group in the full analysis set (FAS).
Overall survival (OS) | Up to approximately 24 months
  Overall survival (OS) is defined as the time between the subject's randomization date and subject's death.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | Up to approximately 24 months
  Progression-free survival (PFS) as assessed by BIRC was defined as the time between the date subjects were randomized and the first observation of disease progression (based on BICR's image-based assessment) or death.
Disease Control Rate (DCR) | Up to approximately 24 months
  Disease Control Rate (DCR) : Percentage of all randomized subjects who rated the best overall response (BOR) as complete response (CR), partial response (PR), and disease stabilization (SD) according to RECIST 1.1 criteria.
Duration of Response (DOR) | Up to approximately 24 months
  Duration of Response (DOR) : defined as the period from the date when tumor response is first recorded to the date when objective tumor progression is first recorded or the date of death.
Treatment Emergent Adverse Event (TEAE) | Up to approximately 24 months
  TEAE is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally emerging, or any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a pre-existing condition during the treatment of BL-B01D1. The type, frequency and severity of TEAE will be evaluated during the treatment of BL-B01D1.
Cmax | Up to approximately 24 months
  Maximum serum concentration (Cmax) of BL-B01D1 will be investigated.
T1/2 | Up to approximately 24 months
  Half-life (T1/2) of BL-B01D1 will be investigated.
Anti-drug antibody (ADA) | Up to approximately 24 months
  Frequency of anti-BL-B01D1 antibody (ADA) will be investigated.

CONTACTS AND LOCATIONS:
Overall Officials: Li Zhang, PHD, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Yang Y, Zhou H, Tang L, Qiu S, Han Y, Ji D, Chen X, Lei F, Qu S, Deng B, Chen L, Huang J, Guo Y, Liu Z, Chen D, Li J, Shu X, Qin Y, Fu Z, Li B, Zhang P, Chen S, Hong J, Wei Y, Qin X, Qu S, Yang K, Lin D, Wang J, Yang L, Xiao S, Zhu H, Zhu Y, Zhang L; BL-B01D1-303 Investigators. Izalontamab brengitecan, an EGFR and HER3 bispecific antibody-drug conjugate, versus chemotherapy in heavily pretreated recurrent or metastatic nasopharyngeal carcinoma: a multicentre, randomised, open-label, phase 3 study in China. Lancet. 2025 Nov 8;406(10516):2235-2243. doi: 10.1016/S0140-6736(25)01954-3. Epub 2025 Oct 19. PMID 41125110